CLINICAL TRIAL: NCT06834217
Title: Characterization and Modulation of Functional Connectivity and Fear Extinction Abnormalities in Obsessive-Compulsive Disorder
Brief Title: Transcranial Direct Current Stimulation and Extinction in Obsessive Compulsive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas Adams, PhD, Associate Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2000039024; R01MH137471 (NIH)
Record Dates: First submitted 2025-01-22; First posted 2025-02-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-06

CONDITIONS: Obsessive Compulsive Disorder (OCD)
Keywords: Anxiety Disorders; Mental Disorders; Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Patients with OCD will be randomized to receive active (real) or sham (placebo) multifocal frontopolar transcranial direct current stimulation (tDCS). All non-clinical controls would not receive any transcranial direct current stimulation (tDCS).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active transcranial direct current stimulation (Active Comparator): Current will be ramped in/out for 30 seconds at the beginning and end of a 20-minute period and a constant current will be delivered for the 20-minutes between ramping.
  Interventions: Device: Active transcranial direct current stimulation
- Sham transcranial direct current stimulation (Sham Comparator): Current will be ramped in and out for 30 seconds followed by a 20-minute period during which no stimulation will be delivered.
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Active transcranial direct current stimulation — Multifocal transcranial direct current stimulation will be delivered. The anode will be placed over the frontal pole (Fpz, 10-20 electroencephalogram [EEG]) and will be surrounded by 5 return electrodes (cathodes). Current will be set at 1.5mA and will be ramped in and out for 30 seconds at the beginning and end of a 20-minute stimulation period.
  Other Names: Transcranial electric stimulation
  Arms: Active transcranial direct current stimulation
Device: Sham transcranial direct current stimulation — Multifocal transcranial direct current stimulation will be delivered. The anode will be placed over the frontal pole (Fpz, 10-20 electroencephalogram [EEG]) and will be surrounded by 5 return electrodes (cathodes). Current will be set at 1.5mA and will be ramped in and out for 30 seconds at the beginning of a 20-minute period.
  Other Names: Placebo transcranial electric stimulation
  Arms: Sham transcranial direct current stimulation

SUMMARY:
Obsessive-compulsive disorder (OCD) is associated with substantial impairments in quality of life and is among the most disabling psychiatric disorders. Exposure therapy is among the first-line of treatments for obsessive-compulsive disorder (OCD) . Extinction learning is thought to be a core mechanism of therapeutic exposure. Fear and safety signal learning are traditionally associated with activity and connectivity within the canonical corticolimbic "fear circuit", which includes the amygdala, medial prefrontal cortex (mPFC), and hippocampus. Transcranial direct current stimulation (tDCS) is a neuromodulation technology that can augment brain plasticity, learning, and memory. The proposed study will test if obsessive-compulsive disorder (OCD) is associated with inhibitory safety learning deficits and if transcranial direct current stimulation (tDCS) normalizes functional connectivity and safety signal processing to recover extinction deficits in obsessive-compulsive disorder (OCD).

DETAILED DESCRIPTION:
The proposed study aims to test if obsessive-compulsive disorder (OCD) is associated with dyconnectivity between the default mode network (DMN) and salience network (SN) (Aim 1), if obsessive-compulsive disorder (OCD) is associated with extinction learning deficits (Aim 2), and if front-polar transcranial direct current stimulation (tDCS) normalizes dysconnectivity and extinction learning in obsessive-compulsive disorder (OCD) (Aim 3).

This study will randomize 180 adults with obsessive-compulsive disorder (OCD) (n=120) and matched non-clinical controls (n=60) for aims 1-3. After providing informed consent, baseline screening, and clinical characterization, participants would complete a three-day experiment. On day 1, all participants would complete structural and resting functional magnetic resonance imaging (fMRI) scans followed by standardized fear conditioning procedures with functional magnetic resonance imaging (fMRI) and measures of fearful responding (i.e., skin conductance response [SCR] and threat expectancy ratings). Participants would be conditioned to two different conditioned stimuli (CS+; CS+A and CS+B) by pairing each CS+ with an aversive shock (unconditioned stimulus [US]) at a 50% schedule of reinforcement. A third, neutral stimulus (CS-), would never be paired with the US. On day 2, participants would complete extinction training for the CS+A, then participants with obsessive-compulsive disorder (OCD) would be randomized (1:1, stratified, double-blind) to receive active or sham multifocal frontopolar transcranial direct current stimulation (tDCS) with resting functional magnetic resonance imaging (fMRI) before, during, and after transcranial direct current stimulation (tDCS). Blocked randomization, stratified by sex, age, and current psychiatric medication usage, would be implemented by an individual who would have no direct contact with the participants and no knowledge of the assignment to the group labels. Participants and assessors will be blind to allocation. All non-clinical controls would not receive any transcranial direct current stimulation (tDCS). Next, extinction training for the CS+B would be completed. On day 3, return of fear testing (spontaneous recovery, context renewal, and reinstatement) would be completed.

Transcranial direct current stimulation (tDCS) would be administered using a battery-driven, Soterix© transcranial electric stimulator. A single anode would be placed over the frontal pole and five return electrodes would be arranged in a circumferential array. Positively charged e-fields produced by this montage would concentrate over the medial frontal pole. Participants in the active-transcranial direct current stimulation (tDCS) condition would receive 20-minutes of offline (while resting with eyes open) frontopolar transcranial direct current stimulation (tDCS) (30-seconds ramp in/out). Participants in the sham-transcranial direct current stimulation (tDCS) condition would receive 30-seconds ramp in/out followed by 20-minutes of no stimulation.

Brain imaging would be performed with a Siemens MAGNETOM Prisma 3T scanner using a 64-channel phased array padded head coil. A vitamin E capsule would be secured to the outer center of the transcranial direct current stimulation (tDCS) anode to create a precise contrast in structural magnetic resonance imaging (MRI). After localization, all participants would undergo anatomical imaging for registration and normalization purposes. 6-min of rs-functional magnetic resonance imaging (fMRI) data would be collected immediately before and after frontopolar transcranial direct current stimulation (tDCS) and four ~5-min blocks rs-functional magnetic resonance imaging (fMRI) sequences would be collected during the 20-min of active- or sham-transcranial direct current stimulation (tDCS) to characterize temporal elements of dosage (e.g., linear change in rs-FC over the time course of transcranial direct current stimulation [tDCS] administration) in exploratory analyses.

ELIGIBILITY:
Inclusion Criteria:

* All Participant Inclusion Criteria would include:

  1. 18 years of age or older
  2. speak English fluently, and
  3. able to provide written and verbal informed consent.
* Obsessive-compulsive disorder (OCD) Inclusion Criteria would include:

  1. meet criteria for OCD as determined by structured clinical interview
  2. exhibit significant current symptoms of OCD
  3. report duration of OCD symptoms of at least 1-year
  4. OCD symptoms are primary or co-primary relative to other psychiatric diagnoses
  5. stable psychiatric treatment (≥8-weeks) or no active treatment.

Exclusion Criteria:

* All Participant Exclusion Criteria would include:

  1. active severe substance use disorder(s)
  2. acute suicidality
  3. history of bipolar or psychotic disorder(s)
  4. significant developmental disabilities
  5. loss of consciousness > 10 minutes
  6. history of traumatic brain injury
  7. major neurological disease
  8. a positive pregnancy test
  9. other brain stimulation or magnetic resonance imaging contraindications
  10. new psychological treatment within the past 8 weeks
  11. active anxiolytic medication use (e.g., benzodiazepine).
* Non-Clinical Control Exclusion Criteria would include:

  1. meet current criteria for a psychiatric disorder as determined by structured clinical interview
  2. active-psychotropic medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Blood oxygen level-dependent (BOLD) response to create functional brain activation maps | Blood oxygen level-dependent (BOLD) will be measured across 3 daily scan sessions separated by ~24 hours each; data will be reported from all 3 sessions.
  Brain activity will be estimated with blood oxygen level-dependent (BOLD) response, which will be measured with magnetic resonance imaging (MRI).
Skin conductance response (SCR) will be measured by collecting electrodermal activity data from the left hand | Skin conductance will be measured across all 3 scan sessions, separated by ~24 hours each; data will be reported from all 3 sessions.
  Skin conductance data will be used as an index of anxious reactivity to experimental cues.
Threat expectancies will be measured by asking participants to rate the probability of receiving a shock using a 0-100 scale with zero equal to 0% chance and 100 equal to 100% chance; higher values are indicative of worse anxious reactivity | Threat expectancies will be assessed at the beginning and end of each of the 3 scan session, separated by ~24-hours each; data will be reported from all 3 sessions.
  Threat expectancies will be used as an index of anxious reactivity to experimental cues.
Functional brain connectivity will be measured blood oxygen level dependent (BOLD) response | Resting functional connectivity will be measured at baseline during first scan session and during transcranial direct current stimulation in the second scan session; scan sessions will be separated by ~24 hours; data from both sessions will be reported.
  Correlations in brain activity between regions and networks measured with blood oxygen level dependent (BOLD) response captured with magnetic resonance imaging (MRI)

CONTACTS AND LOCATIONS:
Locations (1):
- Temple Medical Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw de-identified data will be shared using the National Data Archive.
Time Frame: IPD will be shared within one year of study completion.
Access Criteria: Access to IPD will be public per NDA guidelines.